CLINICAL TRIAL: NCT00133588
Title: Proteomic Profiling for Influenza Vaccination
Brief Title: Proteomic Profiling for Influenza
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-0044
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-05

CONDITIONS: Influenza
Keywords: influenza, vaccine, proteomic profiling, elderly
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Trivalent split Inf

SUMMARY:
The purpose of this study is to evaluate a new method of detecting the flu infection. This method may allow researchers to identify new proteins being made in response to an infection even before symptoms of the infection are present. The goal of this study is not to prevent the flu but to monitor the immune system response. The elderly and those with chronic health problems are at greater risk for complications (i.e., pneumonia, bronchitis [bacterial infection in the lungs], and sinusitis [bacterial infection in the sinuses]) from the flu. Early detection and diagnosis of the flu decreases the number of people with these complications. Participants will include healthy people between the ages of 21-40, between the ages of 60-89, or 90 years and older, who are living in the communities surrounding the 3 study sites in Virginia. There will be 5 study visits, and subjects will participate up to 1 month.

DETAILED DESCRIPTION:
The central hypothesis of this study is that immune responses to vaccination can be quantified by proteomic profiling of serum (and other clinical fluids), and that the host responses to different infectious agents are unique and can be 'fingerprinted' by proteomics. Using influenza virus vaccination, this study proposes to use mass spectrometry platforms to profile and characterize proteins from serum samples obtained from recipients. These samples will be used to develop a proteomic profiling system for monitoring vaccine response and, eventually, early detection/diagnosis of infection. The long-term goal of this approach is to develop tools useful for reducing the morbidity and mortality of influenza from natural and potential bioterrorism-related infections by improving measures of vaccine efficacy and early diagnosis. The primary objective is to use surface-enhanced laser desorption/ionization time-of-flight (SELDI-TOF) mass spectrometry and matrix-assisted laser desorption/ionization time-of-flight (MALDI-TOF) mass spectrometry proteomic profiling tools to analyze a series of serum samples obtained from cohorts of young and elderly subjects, before and after trivalent split-virus influenza vaccination, to identify surrogate markers reflective of the immune response. The secondary objective is to use concurrent T-cell activation, cytokine assays, and hemagglutination inhibition (HI) serologic assays to correlate cellular and humoral responses to influenza vaccination with protein profiling changes. Comparisons of the protein profile data with the T-cell activation, cytokine assays, and HI results will be evaluated using multiple classification algorithms, and potential biomarker proteins will be identified by sequencing with either a MALDI-TOF or electrospray ionization mass spectrometer. Study Participants will include healthy adult volunteers between the ages of 21-40, between the ages of 60-89, or 90 years and older, who are living independently in the communities surrounding the 3 study sites in Virginia. There will be 5 study visits, and subjects will be in the trial for up to 1 month. The primary endpoint of the study is to identify surrogate markers reflective of the immune response and to correlate these markers to cellular and humoral responses (demonstrated with T-cell activation, cytokine assays, and the HI serologic assays) to influenza vaccination. The secondary endpoint is safety. Data on the following solicited local reactions (injection site pain, bruising, redness, tenderness, and induration) and solicited systemic reactions (fever, headache, malaise, myalgia, cough, runny nose, chills, vomiting, arthralgia, rash, and diarrhea) will be collected from Day 0-Day 14 and categorized as none, mild, moderate, and severe. Unsolicited adverse events (including serious adverse events) will be collected and categorized throughout the study by severity, duration, and relatedness to the vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 21 to 40 years of age or between the ages of 60 and 89, or 90 years or older on the day of inclusion.
2. Provides written informed consent.
3. Subject is judged to be healthy on the basis of verbal history.
4. Subject is able to attend scheduled visits and to comply with the study procedures during the entire duration of the study and will be available for 1 month after enrollment.
5. Females of childbearing potential must agree to use contraception and must agree to continue using this method for at least 3 months after enrollment. All females under the age of 60 must have a negative urine pregnancy test at enrollment. Those that have a history of tubal ligation or hysterectomy or are postmenopausal at least 1 year of no menses may be included but must still have a negative urine pregnancy test at enrollment. Acceptable forms of hormonal contraception include the use of oral contraceptives, injectable contraceptives (ie, Depo-ProveraTM) or transdermal contraceptives for a period of 3 months prior to enrollment.
6. Subject must have access to telephone service.

Exclusion Criteria:

1. Subject received an influenza vaccine 6 months preceding enrollment in the study.
2. Subject had physician-diagnosed (preferably by culture) influenza at any time during the past 2 years.
3. Subject had an acute illness with or without fever (temperature greater than or equal to 99.5ºF [oral]) in the 72 hours preceding vaccination.
4. Subject received any vaccine 14 days before enrollment or plans to receive any vaccine during this study.
5. Subject received blood or blood products in the last 3 months.
6. Subject has known or suspected disease(s) of the immune system (ie, rheumatoid arthritis, lupus, lymphoma, human immunodeficiency virus, etc). Stable, controlled osteoarthritis is allowed if medication is only intermittently used for relief of symptoms.

   Subject has underlying unstable chronic disease such as uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg at Visit 1), congestive heart failure, heart attack within the last 6 months, liver, and kidney disease, etc;
7. Subject is currently being treated with an immunosuppressive medications (i.e., cancer therapeutic agents such as Tamoxifen, systemic corticosteroids such as Prednisone, and arthritis medications such as Methotrexate). Please note that inhaled or topical corticosteriods are acceptable.
8. Subject is pregnant or planning to become pregnant within the next 2 months.
9. Subject is breastfeeding.
10. Subject has a history of allergic disease or reactions likely to be exacerbated by any component of the study vaccine, including a history of anaphylaxis or serious vaccine reaction; subject is allergic to eggs, contact lens solution, or has ever had a severe reaction to any influenza vaccine.
11. Subject is allergic to latex rubber;
12. Subject has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. These conditions include, but are not limited to: history of significant renal impairment (dialysis and treatment for kidney disease, including diabetic and hypertensive kidney disease); diabetes mellitus (excluding diet-controlled diabetes); cardiac insufficiency, if heart failure is present (New York Heart Association Functional Class III or IV); arteriosclerotic event during the 2 weeks prior to enrollment (eg, history of myocardial infarction, stroke, recanalization of femoral arteries, or transient ischemic attack); functional or anatomic asplenia; cancer (excluding breast, skin, and prostate cancer diagnosed and treated more than 5 years prior to inclusion).
13. Subject has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
14. Subject has acute respiratory or other active infections or illnesses.
15. Subject has any active neurologic disorders (ie, encephalopathy, optic neuritis/neuropathy, partial facial paralysis, and brachial plexus neuropathy).
16. Subject has a prior history of Guillain-Barré syndrome.
17. Participation in any other interventional drug or vaccine trial within 30 days prior to enrollment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-11; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States